CLINICAL TRIAL: NCT00134797
Title: The Effect of MDRD GFR Reporting on Nephrology Referral Patterns by Internists
Brief Title: Glomerular Filtration Rate (GFR) Reporting on Nephrology Referral Patterns by Internists
Status: Withdrawn | Type: Observational
Why Stopped: PI/study contacts no longer at Institution
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Other Study IDs: CIP #S-04-058
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
Keywords: GFR; serum creatinine
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The addition of an estimate value of glomerular filtration rate (GFR) per Modification of Diet in Renal Disease [MDRD] (LEVEY) equation is being included and reported on all routine chemistry panels in the experimental group. The control group is only having serum creatinine, the current standard of care, reported on routine chemistry panels.

DETAILED DESCRIPTION:
All patients already referred to or being followed by nephrologists were excluded. Inclusion criteria were all patients in the Internal Medicine clinic at NMCSD who were sent to the lab to obtain routine chemistry panels for follow up by their primary care providers. The primary outcome is increased referral to nephrology in accordance with NKF K/DOQI guidelines if GFR values are reported on routine chemistry panels. Key secondary outcomes are Primary Care Provider knowledge of NKF K/DOQI guidelines, specifically when patients with chronic kidney disease need to be referred to a nephrologist for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the Internal Medicine Clinic at Naval Medical Center, San Diego (NMCSD) who were sent to the lab to obtain follow up by their primary care providers.

Exclusion Criteria:

* All patients referred to or being followed by nephrologists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-02; Study Completion 2006-02 (Estimated)

PRIMARY OUTCOMES:
Incraesed referral to nephrology inaccordance with NKF K/DOQI guidelines if GFR values are reported on routine chemistry panels.

SECONDARY OUTCOMES:
Primary Care Provider knowledge of NKF K/DOQI guidelines, specifically when patients with chronic kidney disease need to be referred to a nephrologist for further evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Miller, M.D., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States